CLINICAL TRIAL: NCT05472051
Title: Health and Migration Trajectories of Housekeepers in Bamako: Situation and Acceptability of a Community-based Offer of Sexual Health Services
Brief Title: Health and Migration Trajectories of Housekeepers in Bamako
Acronym: 2DM2K
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 0005s
Record Dates: First submitted 2021-09-13; First posted 2022-07-25 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: HIV Infections; Hepatitis B; Hepatitis C; Tuberculosis; STIs; Sex Behavior
Keywords: Housekeepers; Young girls; Mali; Accès to healthcare; Community-based services
MeSH Terms: conditions — HIV Infections; Hepatitis B; Hepatitis C; Tuberculosis; Sexually Transmitted Diseases; Sexual Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young girls housekeepers: Malian young girls migrating from rural areas towards Bamako to seek for a job as housekeepers. Include young girls aged at least 12 years.
  Interventions: Other: Community-based healthcare offer provided by an the ARCAD Santé PLUS NGO and integrated into the activities of the ADDAD NGO

INTERVENTIONS:
Other: Community-based healthcare offer provided by an the ARCAD Santé PLUS NGO and integrated into the activities of the ADDAD NGO — In the framework of the current activities of the ARCAD Santé PLUS a team formed by a doctor, a nurse and laboratory assistant will provide prevention and medical activities during the community-based activities organized by the housekeepers ADDAD NGO. The medical consultation will propose:
  * HIV screening, including pre- and post- counseling
  * Hepatitis B and hepatitis C screening, including pré- and post- counseling. The HBV vaccine will be proposed to housekeepers with negative results to both HBV and HCV testing
  * Tuberculosis screening will be proposed to housekeepers with symptoms suggesting the possibility of TB
  * For housekeepers sexually active, the medical team will propose a gynecological test in order to screen for genital infections. Furthermore, a pregnancy test will be proposed.
  Medicines for current diseases (headache, diarrhea, etc. will be provided by the medical staff).

SUMMARY:
In Mali, migration from rural zones is a cultural phenomenon existing since 1970. During the dry season (9 months), an important number of young women leave their villages and migrate towards urban zones to seek for a job. In Bamako, the estimated number of housekeepers is 100 000 coming from rural regions and aged between 11 and 19 years. The current healthcare offer seems to be non-adapted to their particularities.

This is a community-based research constructed on the basis of the activities of two NGOs in Mali: ADDAD (association for the defense of the rights of Housekeepers and domestic helpers ) and ARCAD Santé PLUS (the main NGO for healthcare access for HIV, hepatitis, and sexual health services). The research is conducted by the SanteRCom team in the UMR1252 SESSTIM research unit.

The main objective of this observational study is to study the knowledge, beliefs, behaviors and practices in terms of health in general, and sexual health in particular; and to assess the acceptability of an offer of community-based prevention and health services provided by ARCAD Santé PLUS integrated in the activities of ADDAD. The integrating of community-based healthcare offer in a familiar and reassuring framework, such as that of ADDAD, should promote access to health services among housekeepers.

The research is organized in 3 stages:

1. Preliminary qualitative survey based on focus group discussions. Allowing the identification of the housekeepers' needs in terms of prevention and healthcare services; and the behavioral particularities of the housekeepers community. It is planned to conduct 7 focus groups including between 42 and 56 housekeepers.
2. Communication and awareness campaigns in the regions of origin of housekeepers. Campaigns will be constructed on the basis of the results obtained from the preliminary qualitative survey.
3. Communication and awareness campaigns in Bamako; community-based activities for housekeepers will be organized 3 times per week during 5 months by the NGO ADDAD. Activities will include the community-based offer of prevention and healthcare services provided by the NGO ARCAD Santé PLUS, i.e. the novelty in the ADDAD's activities. A quantitative and qualitative surveys will be conducted over 5 months with participants recruited during the community-based activities. It is expected to enroll at least 1134 housekeepers, and to conduct a maximum of 25 individual interviews with selected housekeepers.

ELIGIBILITY:
Inclusion Criteria:

* Being a young girl and working in Bamako as housekeeper
* Speak one of the most current languages : Bambara, Dogon, French
* Being aged at least 12 years,
* To provide written consent. For minors (12 to 17 years old) the consent of a member of the ADDAD NGO as the legal responsible.

Exclusion Criteria:

* Minor housekeepers refusing the presence and signature of the ADDAD's member
* Housekeepers whose mental health would be judged (by the doctor) not appropriate to participate
* Housekeepers not able to understand and/or to sign the written consent

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Young girls working in Bamako as housekeepers (not self-representation)
Study Population: Young girls working in Bamako as Housekeepers being aged at least 12 years.
Sampling Method: Non-Probability Sample
Enrollment: 644 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Acceptability of the community-based offer of healthcare services | 18 month after the start of the study
  Percentage of housekeepers attending the community-based healthcare services during the ADDAD's activities (among the total number of housekeepers attending the ADDAD's activities)
Prevalence of infectious diseases among housekeepers attending the community-based healthcare services and accepting screening | 18 month after the start of the study
  Prevalence of infectious diseases among housekeepers attending the community-based healthcare services and accepting screening:
  Percentage of HIV positive Percentage of HBV positive Percentage of HCV positive Percentage of TB POSITIVE Percentage of genital infectious diseases
Pregnancy | 18 month after the start of the study
  Number of positive pregnancy tests among housekeepers accepting screening
HBV Vaccin | 18 month after the start of the study
  Number of housekeepers accepting HBV vaccine among those negative to both HBV and HCV
Mental health | 18 month after the start of the study
  Prevalence of mental disorders such as depression, anxiety, insomnia, post-traumatic stress

CONTACTS AND LOCATIONS:
Overall Officials: Luis Sagaon Teyssier, PhD, Principal Investigator — UMR 1252 SESSTIM
Locations (1):
- ADDAD, Bamako, Niamakoro, Sièbougouni, Rue 173, Porte 146, Mali